CLINICAL TRIAL: NCT01269307
Title: Combination Ketamine and Propofol vs Propofol for Emergency Department Sedation: A Prospective Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 39736
Record Dates: First submitted 2010-12-10; First posted 2011-01-04 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Sedation
Keywords: Anesthesia; Pain; Procedural sedation; Airway/Anesthesia/Analgesia
MeSH Terms: conditions — Pain | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1:1 ketamine - propofol mixture (Active Comparator)
  Interventions: Procedure: 1:1 ketamine-propofol mixture sedation
- propofol (Active Comparator): propofol
  Interventions: Procedure: Propofol Sedation

INTERVENTIONS:
Procedure: 1:1 ketamine-propofol mixture sedation — Prepare Ketamine and Propofol 10mg/cc of ketamine 10mg/cc of propofol mix 1:1 in 10 or 20 cc syringes Sedation Initial dose 0.05 cc / kg IV bolus. Repeat dose 0.025 - 0.05 every 60-90 seconds as needed to reach and maintain target level of sedation.
  May round to nearest 0.5-1 cc. Note - 1 cc = 5mg of propofol and 5mg of ketamine
  Other Names: Ketofol
  Arms: 1:1 ketamine - propofol mixture
Procedure: Propofol Sedation — Prepare Propofol 10mg/cc of propofol 10 or 20 cc syringes Sedation Initial dose 0.05 cc / kg IV bolus over 30 seconds. Repeat dose 0.025 - 0.05 cc/kg every 30-60 seconds as needed to reach and maintain target level of sedation.
  May round to nearest 0.5 cc Note - 1 cc = 10 mg of propofol
  Other Names: Propofol
  Arms: propofol

SUMMARY:
The purpose of this study is to determine if procedural sedation utilizing a 1:1 mixture of propofol and ketamine is equivalent in complications, patient and physician satisfaction, post-procedure pain level, and procedural outcome to propofol sedation alone.

DETAILED DESCRIPTION:
Procedural sedation (PS) is common in the Emergency Department (ED) for painful or anxiety-producing procedures. In our ED these procedures commonly include fracture and dislocation management and reduction, abscess incision and drainage, lumbar puncture, extensive wound debridement, dilatation and curettage, chest tube placement and cardioversion. Generally a sedative-hypnotic agent is combined with an analgesic in order to provide this sedation. The ideal agents to utilize remain unclear. The ED environment is substantially different than the operative suite or many outpatient areas and literature from these areas has limited applicability.

In many ED's, including our own, propofol combined with either a short acting or long acting narcotic has become very commonly utilized. Propofol has many advantages including rapid onset, rapid recovery, strong sedative and amnestic properties, and euphoric effects. However like many sedative-hypnotics it possesses strong respiratory depressive properties and has cardio-depressant and vasodilatation effects that can lead to hypotension. These effects can be potentiated by concomitant narcotic administration as opioid agonists posses similar properties.2

ED literature on complications associated with propofol sedation is variable, secondary to significant differences in rapidity of administration of the medication, the type of analgesic provided, the definitions of complications, the amount of pre-oxygenation provided, and the variability in experience of medical providers. Most literature suggests that the overall rate of sub-clinical respiratory depression, measured by indicators such as end-tidal CO2 changes, is approximately 30-40% of patients1-3. The clinical importance of these changes is unclear. Clinical respiratory depression, measure by hypoxemia, need for verbal or tactile stimulation, bag valve mask ventilation (BVM), and airway positioning, is reported in 1-25% of patients, with the need for BVM ranging from 0-4.6% of patients1-6. It is noteworthy that one study, utilizing a slow infusion rate and only long-acting narcotics administered greater than 20 minutes prior to the start of sedation, prospectively demonstrated only a 0.88% rate of hypoxemia and a 0% rate of BVM while maintaining a similar total average dose, patient satisfaction, and successful outcome6. However this has not been replicated, and the data from other ED studies seems to suggest rates of clinical respiratory depression of 10-12% with BVM use averaging 4%1-6. The only clear conclusion to be drawn from the medical literature in this regard is that some respiratory depression and need for airway management can occur, but the rate is likely heavily dependent on exact protocols and definitions, make comparison between centers and studies difficult.

Because of interest in developing effective sedation regimens that might mitigate some of the complications of propofol plus narcotic regimens (hereafter termed propofol sedation), a technique of combining propofol and ketamine has been described for use in the ED. This combination is long-standing in some settings 7-10 and its use in the ED has been described 9,12,13. Ketamine is a dissociative hypnotic that acts by binding N-methyl-D-aspartate (NMDA) receptors, blocking their excitatory function. It has analgesic, amnestic, and dissociative, effects 9-12. It has the beneficial properties of maintaining respiratory drive, maintaining muscular airway control while still providing pain relief and dissociation. Its use as a single agent for ED sedation in adults has been limited by concern about dysphoria at anesthetic doses as well as post-sedation nausea and vomiting. It can also cause tachycardia and hypertension. However the intuitive off-setting of the somewhat opposite side effects of propofol and ketamine have created significant interest in sedation regimens utilizing both agents. (ie propofol decrease heart rate (HR), blood pressure (BP), respiratory drive and airway maintenance, is euphoric and is an anti-emetic. Ketamine increases HR, BP and increases or maintains respiratory drive and airway maintenance, but is dysphoric and can be nauseating.) An ED study was published in 2007 describing the use of a fixed dose mixture of 1:1 propofol and ketamine (also termed "Ketofol") in a single syringe, allowing for easy dose titration 12. This study showed high patient and physician satisfaction (mean of 10 on a 1-10 scale), high rates of procedural success, and an extremely low rate of complications (2.5% rate of hypoxemia, 0.9% rate of BVM ventilation)12. Another study, in children with different dosing parameters, recently suggested a similarly low rate of BVM (0%) but a higher rate of respiratory depression (15%)13. Interestingly this study used a lower amount of ketamine and higher dose of propofol, which perhaps contributed to the increased rate of respiratory depression. Retrospective data from our use of fixed dose 1:1 ketamine and propofol demonstrates a similar safety profile with 7% of patients having some respiratory depression or requiring airway management and an absolute rate of 2% requiring BVM. We have commonly used this combination in our ED since 2007.

Currently in our ED both propofol sedation and ketamine plus propofol sedation are variably employed, depending mainly on prescriber preference. Because the literature has significant variability in the reported complication rates of the two regimens, no firm conclusion is possible about the relative equivalence or superiority of one regimen compared to the other. Attending physician preference currently dictates the choice of an agent for our patients in lieu of any robust evidence to guide our selection. Further, there is no data to measure the relative patient satisfaction and provider ease of utilization of either of these regimens, important factors in the selection of sedation agents.

We plan to conduct a prospective, randomized, equivalence trial of a fixed ratio of 1:1 ketamine and propofol vs propofol alone sedation. We will measure sub-clinical and clinical respiratory depression, the need for active airway management, unpleasant complications such as post-sedation nausea and vomiting, dysphoria and emergence reactions, patient and provider satisfaction, and post-procedure and follow up pain.

ELIGIBILITY:
Inclusion Criteria:

* English speaking patients eighteen and older who present to the University of Utah Emergency Department and require, in their treating physician's opinion, procedural sedation for a procedure or radiologic study performed in the Emergency Department.

Exclusion Criteria:

* Include prior sensitization or allergic reaction to propofol, ketamine, soy or egg products; hemodynamic instability; clinical evidence of head injury, increased intracranial or intraocular pressure; use of drugs known to interact with either study agent, pregnancy with a live intra-uterine pregnancy (i.e. undergoing Dilation and Curettage for intrauterine fetal demise or spontaneous abortion is not an exclusion criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
airway complications | within 12 months of study completion
  The use of any: Adjunctive airway device (nasopharyngeal airway (NPA)/oropharyngeal airway (OPA), Jaw thrust or other airway maneuver., Use of Bag Valve Mask (BVM) for ventilation and reversal medications (i.e. Narcan).
subclinical respiratory depression | within 12 months of study completion
  subclinical respiratory depression (hypoxemia despite supplemental oxygen noted on pulse-oximetry, loss of End-tidal carbon dioxide concentration in the expired air (ETCO2) waveform for 15 seconds or greater, systolic pressure (SBP) below 80mm Hg, cardiac arrhythmias.)
satisfaction | within 12 months of study completion
  Following sedation, questionnaires were completed by the sedating physician, any consultant physician, nurse, and patient

CONTACTS AND LOCATIONS:
Overall Officials: Scott Youngquist, MD MSc, Principal Investigator — University of Utah; Virgil Davis, MD, Principal Investigator — University of Utah; Troy Madsen, MD, Principal Investigator — University of Utah; Anas Sawas, MS MPH, Principal Investigator — University of Utah; Matthew Ahern, DO, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Miner JR, Danahy M, Moch A, Biros M. Randomized clinical trial of etomidate versus propofol for procedural sedation in the emergency department. Ann Emerg Med. 2007 Jan;49(1):15-22. doi: 10.1016/j.annemergmed.2006.06.042. Epub 2006 Sep 25. PMID 16997421
- [Background] Miner JR, Gray RO, Stephens D, Biros MH. Randomized clinical trial of propofol with and without alfentanil for deep procedural sedation in the emergency department. Acad Emerg Med. 2009 Sep;16(9):825-34. doi: 10.1111/j.1553-2712.2009.00487.x. PMID 19845550
- [Background] Burton JH, Miner JR, Shipley ER, Strout TD, Becker C, Thode HC Jr. Propofol for emergency department procedural sedation and analgesia: a tale of three centers. Acad Emerg Med. 2006 Jan;13(1):24-30. doi: 10.1197/j.aem.2005.08.011. Epub 2005 Dec 19. PMID 16365337
- [Background] Zed PJ, Abu-Laban RB, Chan WW, Harrison DW. Efficacy, safety and patient satisfaction of propofol for procedural sedation and analgesia in the emergency department: a prospective study. CJEM. 2007 Nov;9(6):421-7. doi: 10.1017/s148180350001544x. PMID 18072987
- [Background] Friedberg BL. Propofol-ketamine technique: dissociative anesthesia for office surgery (a 5-year review of 1264 cases). Aesthetic Plast Surg. 1999 Jan-Feb;23(1):70-5. doi: 10.1007/s002669900245. PMID 10022941
- [Background] Friedberg BL. Propofol ketamine anesthesia for cosmetic surgery in the office suite. Int Anesthesiol Clin. 2003 Spring;41(2):39-50. doi: 10.1097/00004311-200341020-00006. No abstract available. PMID 12711912
- [Background] Messenger DW, Murray HE, Dungey PE, van Vlymen J, Sivilotti ML. Subdissociative-dose ketamine versus fentanyl for analgesia during propofol procedural sedation: a randomized clinical trial. Acad Emerg Med. 2008 Oct;15(10):877-86. doi: 10.1111/j.1553-2712.2008.00219.x. Epub 2008 Aug 27. PMID 18754820
- [Background] Slavik VC, Zed PJ. Combination ketamine and propofol for procedural sedation and analgesia. Pharmacotherapy. 2007 Nov;27(11):1588-98. doi: 10.1592/phco.27.11.1588. PMID 17963466
- [Background] Bowdle TA, Radant AD, Cowley DS, Kharasch ED, Strassman RJ, Roy-Byrne PP. Psychedelic effects of ketamine in healthy volunteers: relationship to steady-state plasma concentrations. Anesthesiology. 1998 Jan;88(1):82-8. doi: 10.1097/00000542-199801000-00015. PMID 9447860
- [Background] Willman EV, Andolfatto G. A prospective evaluation of "ketofol" (ketamine/propofol combination) for procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2007 Jan;49(1):23-30. doi: 10.1016/j.annemergmed.2006.08.002. Epub 2006 Oct 23. PMID 17059854
- [Background] Sharieff GQ, Trocinski DR, Kanegaye JT, Fisher B, Harley JR. Ketamine-propofol combination sedation for fracture reduction in the pediatric emergency department. Pediatr Emerg Care. 2007 Dec;23(12):881-4. doi: 10.1097/pec.0b013e31815c9df6. PMID 18091596